CLINICAL TRIAL: NCT06374095
Title: Basiliximab With One Day or Seven Days RATG Induction Therapy in Renal Transplantation: a Matched-cohort Observational Study
Brief Title: 1 vs 7 RATG Infusions in Renal Transplantation
Acronym: ONSET
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: ONSET
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Kidney Replacement
Keywords: Kidney transplant; Basiliximab; RATG induction therapy
MeSH Terms: interventions — thymoglobulin; Basiliximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 25 consecutive recipients of a single or dual kidney transplant from ideal or marginal donors who, from 01/04/2023 to 31/12/2023, were induced with one single perioperative RATG infusion (Patients) at the Renal Transplant Center of the Azienda Socio Sanitaria Territoriale (ASST) of the Papa Giovanni XXIII Hospital, in Bergamo (Italy)
  Interventions: Drug: RATG; Drug: Basiliximab
- Reference patients: The most recent 50 consecutive recipients (Reference-Patients) of a single or dual kidney transplant from ideal or marginal donors who before 01/04/2023 were induced with seven perioperative RATG infusions (on top of the same induction and maintenance treatment used for patients receiving one single RATG infusion) at the Renal Transplant Center of the (ASST) of the Papa Giovanni XXIII Hospital, in Bergamo (Italy)
  Interventions: Drug: RATG; Drug: Basiliximab

INTERVENTIONS:
Drug: RATG — Thymoglobulin, Genzyme corporation, Italy.
  Other Names: Thymoglobulin
Drug: Basiliximab — Simulect, Novartis, Italy.
  Other Names: Simulect

SUMMARY:
This trial is to compare the risk/benefit profile over six-month follow-up of two induction immunosuppressive regimens based on one or seven low-dose perioperative RATG infusions on top of the same induction therapy with basiliximab and steroid (progressively tapered post-transplant) and maintenance therapy with calcineurin inhibitors and mycophenolate mofetil/mycophenolic acid in 75 recipients (25 Patients and 50 Reference-Patients) of a single or dual first kidney transplant from an ideal or marginal donor at a single Renal Transplant Center.

DETAILED DESCRIPTION:
In patients receiving a kidney transplant, it is necessary to use immunosuppressive drugs that serve to reduce or prevent the risk of rejection. Some of these drugs are infused only in the first days of the transplant to more effectively reduce the reactivity of the immune system when the risk of rejection is highest. Among these are thymoglobulins, antibodies that destroy immune system cells (lymphocytes) which can cause rejection. For this reason, in their Center the investigators have developed a protocol that provides for the infusion of thymoglobulins for seven consecutive days starting from the day of the transplant. The first infusion begins even before the transplant is performed so that the lymphocytes are destroyed before the kidney is implanted and can therefore be recognized by the immune system as a foreign organ. This first administration is therefore certainly the most important, to the point that perhaps subsequent infusions of thymoglobulins may not even be necessary. Based on this reasoning, starting from April 1st 2023 the investigators began to infuse only the first dose of thymoglobulins, always starting the infusion before the transplant was performed, avoiding subsequent administrations. The goal was to maintain the same anti-rejection efficacy, but reducing the risk of side effects. In fact, thymoglobulins reduce the number of white blood cells and platelets in the blood and can increase the risk of opportunistic infections which are facilitated by the fact that the activity of the immune system is reduced by thymoglobulins. In other words, the effects of thymoglobulins on the immune system that serve to reduce the risk of rejection are the same as those that increase the risk of infections.

At this point the investigators would therefore like to verify whether actually infusing a single dose of thymoglobulin starting before the transplant can maintain the same anti-rejection effect that is obtained by administering seven doses of thymoglobulin, while reducing the risk of side effects. For this reason, in this study they want to compare the data already collected for clinical reasons in kidney transplant recipients treated with a single dose of thymoglobulin with the data, also already collected, in kidney transplant recipients who instead received all seven doses of thymoglobulin. The latter must have the same characteristics as patients who have received a single dose of thymoglobulins. In essence the investigators should compare two groups of patients who are very similar in terms of the type of transplant performed (for example single or double) and the other anti-rejection therapies administered in addition to thymoglobulins and who differ only in having received one or seven infusions. All patients will have received the transplant from the same surgical team and will have been monitored and treated by the same nephrology team based on the same standardized clinical monitoring and immunosuppressive treatment protocols (regardless of the number of thymoglobulin doses). In this way, any differences in the risk of rejection or side effects that may emerge between the two groups could only be explained by the difference in treatment with thymoglobulins (with a single dose or with seven doses).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive recipients of a single or dual kidney transplant from ideal or marginal donors who, from 01/04/2023 to 31/12/2023, were induced with one single perioperative RATG infusion
* Consecutive recipients (Reference-Patients) of a single or dual kidney transplant from ideal or marginal donors who before 01/04/2023 were induced with seven perioperative RATG infusions (on top of the same induction and maintenance treatment used for patients receiving one single RATG infusion)

Exclusion Criteria:

* Living donor recipients, second transplant recipients or patients receiving a multiorgan transplant, and patients with a peak panel reactive antibody titer >30% or positive B cell cross-match

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive recipients of a single or dual kidney transplant from ideal or marginal donors at the Renal Transplant Center of the Azienda Socio Sanitaria Territoriale (ASST) of the Papa Giovanni XXIII Hospital, in Bergamo (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of thrombocytopenia and/or leukopenia | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Incidence of thrombocytopenia and/or leukopenia requiring or not requiring down-titration or transient withdrawal of mycophenolate mofetil/ mycophenolic acid (and/or RATG)

SECONDARY OUTCOMES:
Occurrence of anemia | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Occurrence of anemia requiring treatment with erythropoiesis stimulating agents
Occurrence of viral infections | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Polyomavirus BK (BKV) and/or Cytomegalovirus (CMV) infection/reactivations
Occurrence of pneumonia | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Pneumocystis carinii pneumonia
Occurrence of opportunistic infections | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Systemic candidiasis and any other opportunistic infection
Occurrence of delayed graft function | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Delayed Graft Function defined as need of dialysis during the first week post-transplant
Occurrence of allograft rejection | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Acute allograft rejection (overall, steroid-resistant and biopsy-proven rejections considered separately)
Occurrence of biopsy proven rejection | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Banff score for biopsy proven rejections
Survival | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Six-month patient/graft survival
Platelet and WBC counts | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Six-month time course of platelet and WBC counts
Creatinine levels | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Six-month time course of serum creatinine levels
Adverse events | From day 0 post-transplant up to 10 days or patient discharge, then at 2, 3 and 4 weeks post-transplant and every 1 month up to 12 months
  Incidence of serious and non-serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- ASST HPG23 - Unità di Nefrologia, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebranchu Y, Bridoux F, Buchler M, Le Meur Y, Etienne I, Toupance O, Hurault de Ligny B, Touchard G, Moulin B, Le Pogamp P, Reigneau O, Guignard M, Rifle G. Immunoprophylaxis with basiliximab compared with antithymocyte globulin in renal transplant patients receiving MMF-containing triple therapy. Am J Transplant. 2002 Jan;2(1):48-56. doi: 10.1034/j.1600-6143.2002.020109.x. PMID 12095056
- [Background] Remuzzi G, Lesti M, Gotti E, Ganeva M, Dimitrov BD, Ene-Iordache B, Gherardi G, Donati D, Salvadori M, Sandrini S, Valente U, Segoloni G, Mourad G, Federico S, Rigotti P, Sparacino V, Bosmans JL, Perico N, Ruggenenti P. Mycophenolate mofetil versus azathioprine for prevention of acute rejection in renal transplantation (MYSS): a randomised trial. Lancet. 2004 Aug 7-13;364(9433):503-12. doi: 10.1016/S0140-6736(04)16808-6. PMID 15302193
- [Background] Thiyagarajan UM, Ponnuswamy A, Bagul A. Thymoglobulin and its use in renal transplantation: a review. Am J Nephrol. 2013;37(6):586-601. doi: 10.1159/000351643. Epub 2013 Jun 12. PMID 23774740